CLINICAL TRIAL: NCT06598618
Title: Compare the Effects of Instrument Assisted Soft Tissue Mobilization (IASTM) and Muscle Energy Technique on Iliotibial Band Tightness in Patients With Patellofemoral Syndrome.
Brief Title: Comparison of IASTM and Muscle Energy Technique in Patellofemoral Pain Syndrome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01872 Aleezae Shamim
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: IASTM; MET; iliotibial band; patellofemoral pain syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graston technique+ Conventional PT (Active Comparator)
  Interventions: Other: Graston technique+ Conventional PT
- Muscle energy technique + Conventional PT (Other)
  Interventions: Other: Muscle energy technique + Conventional PT

INTERVENTIONS:
Other: Graston technique+ Conventional PT — IASTM technique (graston technique) on iliotibial band. Frequency 2 sessions of stroking with 20 seconds rest in between 3 times/week for 3 consecutive weeks Intensity as tolerated by patient. Conventional PT including 1- Therapeutic ultrasound at frequency of 3.5 MHZ for 10 minutes. 2- Stretching exercise of hamstrings. 3-Isometric exercises of Quadriceps
  Arms: Graston technique+ Conventional PT
Other: Muscle energy technique + Conventional PT — Muscle energy technique (post facilitation stretch) on iliotibial band. Frequency 10 repetitions 3 times/week for 3 consecutive weeks Intensity starting from 50 percent resistance across barrier provided by physiotherapist.. Conventional PT including 1- Therapeutic ultrasound at frequency of 3.5 MHZ for 10 minutes. 2- Stretching exercise of hamstrings. 3-Isometric exercises of Quadriceps.
  Arms: Muscle energy technique + Conventional PT

SUMMARY:
The aim of this randomized controlled trial is to compare the effect of Instrument Assisted Soft Tissue Mobilization (IASTM) and muscle energy technique on iliotibial band tightness on pain, range of motion and functional mobility in patients with patellofemoral pain syndrome.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) is termed as anterior knee pain and is characterized by peripatellar or retro patellar pain as a result of changes in the physical and biochemical components of the patellofemoral joint due to increased load during activities such as running, squatting, going up and down stairs, cycling and jumping. Patellofemoral syndrome is one of the most common knee conditions seen by clinicians. In active individuals, it may account for 25% to 40% of all knee problems The iliotibial band is a lateral thickening of the fascia which attaches to the tensor fascia lata proximally. Most of the lateral retinaculum (superficial oblique and deep transverse portion) arises from the ITB, therefore the ITB indirectly provides lateral stabilisation and acts as a passive restraint to medial patella glide. A tight ITB could theoretically lead to lateral patella tracking, lateral patella tilt and lateral patella compression. Several authors have suggested that tightness in the iliotibial band may contribute to patellofemoral syndrome and knee pain by pulling the patella laterally, thereby causing abnormal tracking of the patella in the trochlear groove.

The Instrument-Assisted Soft Tissue Mobilization (IASTM) technique is the most frequent soft tissue mobilization techniques. It involves the use of a tool that causes mechanical micro-traumatic injury to the treated area. As a result, an inflammatory reaction is elicited, speeding up the healing process and restoring the flexibility and integrity of the tissue and cartilage healing. The therapeutic effects of this approach appear to include decreasing tissue adhesion, enhancing the number of fibroblasts, and stimulating collagen synthesis.

Muscle energy technique is a soft tissue technique designed to improve musculoskeletal function through stretching tight muscles and fascia, to reduce pain and improve circulation. MET is characterized by a patient-induced skeletal muscle contraction against physiotherapist resistance in a controlled direction and position. The pathological barrier of a muscle is located through joint positioning which is followed by active muscle contraction by the patient moving away from the resistance followed by relaxation of the muscle. A new pathological barrier is located through passive movement and the process is repeated.

The rationale for the use of these techniques is to compare the effects of IASTM and MET of iliotibial band tightness in improving pain, range of motion and functional mobility in patients with patellofemoral pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* • Age between 18 and 35 years

  * Both Genders.
  * Anterior or retro patellar knee pain for at least the past 3 months.
  * Knee pain during at least 3 of the following activities: ascending/descending stairs, squatting, hopping/ running, and prolonged sitting.
  * Retro patellar pain in patellar grind test (positive clarke's sign).
  * A score of at least 3 on the visual analog scale (VAS).
  * Positive Ober's test.

Exclusion Criteria:

* • Any meniscal or ligament tears of knee.

  * Knee osteoarthritis.
  * Any previous surgery of lower limb.
  * Patellar fracture or fracture of lower extremity.
  * Having received knee injections of corticosteroids or hyaluronic acid.
  * Osteoporosis of knee joint.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-09-28 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 3 weeks
  The VAS is a reliable, valid, responsive, and frequently used pain outcome measure. It consists of a bidirectional 10 cm straight line with two labels, that is, "no pain" and "worst possible pain", located at either end of the line.
  VAS consists of a bidirectional 10 cm straight line with two labels, that is, "no pain" and "worst possible pain", located at either end of the line. Patients are instructed to draw a vertical mark on the line indicating their pain level.
Goniometer | 3 weeks
  A goniometer is an instrument that measures the available range of motion at a joint.
Kujala questionnaire | 3 weeks
  The Kujala AKPS is a 13-item screening instrument designed to assess Patellofemoral pain in adolescents and young adults. The total score of the questionnaire is equal to 100, which shows the maximum function of the knee joint.

CONTACTS AND LOCATIONS:
Overall Officials: KINZA ANWAR, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No